CLINICAL TRIAL: NCT06729099
Title: Validity of Brain Metastasis Risk Predictive Model in Hormone Positive Breast Cancer Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Moheb Ibrahim Melek, Clinical oncology specialist, Assiut University
Other Study IDs: Predictive model
Record Dates: First submitted 2024-12-08; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer, Estrogen Receptor-Positive
Keywords: breast cancer; Hormonal receptor positive; brain metastasis risk; Prediction model
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Low-risk group: Brain metastasis risk prediction model score 0-4 points.
- Medium-risk group: Brain metastasis risk prediction model score 5-10 points.
- High-risk group: Brain metastasis risk prediction model score >10 points.

SUMMARY:
This study aims to validate a prediction model of brain metastasis risk for females with HR+ breast cancer by using variables collected at diagnosis.

DETAILED DESCRIPTION:
1. Data collection:

   Age at BC diagnosis, tumor size, axillary adenopathy, clinical stage, HER2 status, Ki67 proliferation index and the modified Scarff-Bloom-Richardson grade of differentiation.
2. Analysis Plan:

   Continuous variables as means and standard deviation (SD) if they follow a normal distribution; if not, as medians and IQR (interquartile range). Numbers and percentages display categorical variables.
3. Model validation:

The association between covariates and the diagnosis of brain metastases by performing logistic regression analyses; odds ratio (OR), 95 % confidence intervals (CI), and p-value will be estimated. Variables with a p-value < 0.05 in the univariate logistic regression analysis will be further assessed in a multivariate logistic regression analysis.

For the clinical use of the model, we will use a score to each variable as that designed by Cacho-Díaz B. et. al. then, we will categorize patients into three risk groups according to the sum of the scores. We will employe a Cox regression analysis to assess each group's risk of developing brain metastases. Adjusted hazard ratios (aHRs), 95 % CIs, and p values will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of HR-positive primary invasive breast cancer.

Exclusion Criteria:

1. Patients if they were diagnosed with brain metastases at the time of initial breast cancer diagnosis or within the subsequent three months.
2. Bilateral breast cancer.
3. Synchronic cancer (i.e., lung cancer, melanoma).
4. Paitents presenting neurologic symptoms without follow-up or lacking a contrast-enhanced magnetic resonance image (cMRI).
5. Incomplete clinicopathological information at the time of diagnosis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical records of women with HR+ breast cancer in clinical oncology department in Assiut University Hospital, Assiut, Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Validity of prediction model of brain metastases risk for females with HR+ breast cancer | 2 years
  A Cox regression analysis to assess each group's risk of developing brain metastases. Adjusted hazard ratios (aHRs), 95 % CIs, and p values will be evaluated.

IPD SHARING:
Plan to Share IPD: Undecided
Not yet decided.